CLINICAL TRIAL: NCT00068510
Title: Phase I Dose Escalation Study of Autologous Tumor Lysate-Pulsed Dendritic Cell Immunotherapy for Malignant Gliomas
Brief Title: Vaccine Therapy in Treating Patients With Malignant Glioma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000327711; UCLA-0304053
Record Dates: First submitted 2003-09-10; First posted 2003-09-11 (Estimated); Last update posted 2020-08-03 (Actual); Status verified 2013-08

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: adult glioblastoma; adult anaplastic astrocytoma; adult brain tumor; adult giant cell glioblastoma; adult gliosarcoma; adult anaplastic oligodendroglioma
MeSH Terms: conditions — Central Nervous System Neoplasms; Glioblastoma; Astrocytoma; Brain Neoplasms; Gliosarcoma; Oligodendroglioma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- autologous tumor lysate-pulsed DC (Experimental)
  Interventions: Biological: therapeutic autologous dendritic cells

INTERVENTIONS:
Biological: therapeutic autologous dendritic cells

SUMMARY:
RATIONALE: Vaccines made from a person's white blood cells mixed with tumor proteins may make the body build an immune response to kill tumor cells.

PURPOSE: This phase I trial is studying the side effects and best dose of vaccine therapy in treating patients with malignant glioma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the dose-limiting toxicity and maximum tolerated dose of autologous tumor lysate-pulsed dendritic cells in patients with malignant gliomas.
* Determine survival, tumor progression, and cellular immune response in patients treated with this regimen.

OUTLINE: This is a dose-escalation study.

Patients undergo leukapheresis for the collection of peripheral blood mononuclear cells (PBMC). Autologous dendritic cells (DC) are prepared from autologous PBMC exposed to sargramostim (GM-CSF) and interleukin-4 and pulsed with autologous tumor lysate. Patients receive autologous tumor lysate-pulsed DC intradermally on days 0, 14, and 28 in the absence of unacceptable toxicity.

Cohorts of 6-12 patients receive escalating doses of autologous tumor lysate-pulsed DC until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

Patients are followed every 2 months for 2 years.

PROJECTED ACCRUAL: A total of 3-18 patients will be accrued for this study within 9-18 months.

ELIGIBILITY:
Eligibility Criteria:

* Histologically confirmed diagnosis of one of the following malignant gliomas:
* Anaplastic astrocytoma
* Glioblastoma multiforme
* Anaplastic oligodendroglioma
* Malignant mixed oligoastrocytoma
* WHO grade III or IV disease
* Newly diagnosed disease
* Bidimensionally measurable disease by contrast-enhancing MRI
* Surgically accessible tumor for which resection is indicated
* Previously treated with or plan to undergo treatment with conventional external beam radiotherapy
* Age 18 and over
* Performance status Karnofsky 60-100%
* Life expectancy at least 8 weeks
* Hemoglobin at least 10 g/dL
* Absolute granulocyte count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* SGOT and SGPT no greater than 2 times normal
* Alkaline phosphatase no greater than 2 times normal
* Bilirubin no greater than 1.5 mg/dL
* Hepatitis B negative
* Hepatitis C negative
* BUN no greater than 1.5 times normal
* Creatinine no greater than 1.5 times normal
* HIV negative
* Syphilis serology negative
* Afebrile
* Negative pregnancy test
* Fertile patients must use effective contraception
* At least 2 weeks since prior chemotherapy (6 weeks for nitrosoureas) and recovered.
* At least 2 weeks since prior corticosteroids
* At least 2 weeks since prior radiotherapy and recovered
* More than 72 hours since prior systemic antibiotics

Exclusion Criteria:

* active infection
* immunodeficiency
* autoimmune disease that may be exacerbated by immunotherapy, including any of the following:
* Rheumatoid arthritis
* Systemic lupus erythematosus
* Vasculitis
* Polymyositis-dermatomyositis
* Scleroderma
* Multiple sclerosis
* Juvenile-onset insulin-dependent diabetes
* allergy to study agents
* pregnant or nursing
* underlying condition that would contraindicate study therapy
* concurrent severe or unstable medical condition that would preclude giving informed consent
* psychiatric condition that would preclude study participation or giving informed consent
* other malignancy within the past 5 years except adequately treated basal cell or squamous cell skin cancer, localized prostate cancer, or carcinoma in situ of the cervix
* concurrent chemotherapy during and for 2 weeks after administration of study vaccine
* concurrent corticosteroids prior organ allograft
* antihistamine therapy within 5 days before or after administration of study vaccine
* other concurrent investigational agents
* concurrent adjuvant therapy during and for 2 weeks after administration of study vaccine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2003-06; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Dose Limiting Toxicity | 4 weeks

SECONDARY OUTCOMES:
Time to tumor progression, overall survival and cellular immune responses in brain tumor patients injected with tumor lysate pulsed dendritic cells | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Linda M. Liau, MD, PhD, Principal Investigator — Jonsson Comprehensive Cancer Center
Locations (1):
- Jonsson Comprehensive Cancer Center at UCLA, Los Angeles, California, United States

REFERENCES:
- [Result] Liau LM, Prins RM, Kiertscher SM, Odesa SK, Kremen TJ, Giovannone AJ, Lin JW, Chute DJ, Mischel PS, Cloughesy TF, Roth MD. Dendritic cell vaccination in glioblastoma patients induces systemic and intracranial T-cell responses modulated by the local central nervous system tumor microenvironment. Clin Cancer Res. 2005 Aug 1;11(15):5515-25. doi: 10.1158/1078-0432.CCR-05-0464. PMID 16061868
- [Derived] Prins RM, Wang X, Soto H, Young E, Lisiero DN, Fong B, Everson R, Yong WH, Lai A, Li G, Cloughesy TF, Liau LM. Comparison of glioma-associated antigen peptide-loaded versus autologous tumor lysate-loaded dendritic cell vaccination in malignant glioma patients. J Immunother. 2013 Feb;36(2):152-7. doi: 10.1097/CJI.0b013e3182811ae4. PMID 23377664